CLINICAL TRIAL: NCT07043023
Title: LIDOCRIT : Effect of Continuous Intravenous LIDOcaine on Discomfort in Postoperative CRITical Care Inpatients
Acronym: LIDOCRIT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 35RC22_8943_LIDOCRIT; 2024-517749-15-00 (EU CTIS Number); 25.00870.000409 (Other: CPP)
Record Dates: First submitted 2025-06-13; First posted 2025-06-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Post-surgery Critical Incare
Keywords: critical incare; post-surgery; lidocaine; placebo
MeSH Terms: interventions — Lidocaine; Pharmaceutical Preparations; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, multicentre, double-blind, placebo-controlled clinical trial. Comparison of Lidocaine IVSE to placebo. Randomisation by block in 1:1, stratified according to centre.
  All patients were randomised as soon as possible and within 6 hours of leaving the operating theatre, into one of two groups:
  * Experimental group: 2% Lidocaine, bolus of 0.075 ml/kg of real weight (i.e. 1.5 mg/kg) then IVSE at 0.05 ml/kg/h (i.e. 1 mg/kg/h) for 48 hours.
  * Control group: placebo (sodium chloride 0.9%), bolus of 0.075 ml/kg real weight then IVSE at 0.05 ml/kg/h for 48 hours Treatment is started as soon as possible, up to 2 hours after randomisation. The syringes were prepared by a 'friendly' service (not involved in patient follow-up) and were of identical size to maintain blindness. The randomisation arm was not known to the doctor in charge of the patient.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The syringes are prepared by a 'friendly' service (not involved in the patient's follow-up) and are of identical format whatever the experimental treatment, in order to maintain blindness. The randomisation arm is not known to the doctor in charge of the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): Lidocaine 2%, bolus of 0.075 ml/kg real weight (i.e. 1.5 mg/kg) then continuous intravenous administration by electric syringe at 0.05 ml/kg/h (i.e. 1 mg/kg/h) for 48 hours
  Interventions: Drug: Lidocaine (drug)
- Placebo (Placebo Comparator): Placebo (sodium chloride 0.9%), bolus of 0.075 ml/kg of real weight then continuous intravenous administration by electric syringe at 0.05 ml/kg/h for 48h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine (drug) — Lidocaine 2%, bolus of 0.075 ml/kg real weight (i.e. 1.5 mg/kg) then IVSE at 0.05 ml/kg/h (i.e. 1 mg/kg/h) for 48 hours
  Other Names: Lidocaine 2%
  Arms: Lidocaine
Drug: Placebo — Placebo (sodium chloride 0.9%), bolus of 0.075 ml/kg of real weight then IVSE at 0.05 ml/kg/h for 48h
  Other Names: Sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
Although pain management in intensive care units and intensive care units has improved since the DOLOREA study, research into therapies and techniques to optimise analgesia is still needed. The many adverse effects of morphine are well known, and it has been observed that excessive sedation during the first 48 hours is associated with an increase in mortality and length of stay. Multimodal analgesia protocols, preferably including non-morphine analgesics, could improve the comfort of critical care patients.

Comfort is a central element of critical care and perioperative management, as demonstrated by Patients-Reported Outcomes (PRO), new assessment tools that take into account the patient as a whole. The (Inconfort of REAnimation Patients) IPREA questionnaire, a specific scale for assessing the comfort of critical care patients, is an example of a PRO.

Lidocaine is a voltage-dependent sodium channel blocker, used as a local anaesthetic and antiarrhythmic agent, whose intravenous administration produces analgesic effects, particularly on hyperalgesia. The widely demonstrated clinical benefits in scheduled and major surgery (reduced post-operative pain, reduced doses of anaesthetic agents and opiates, reduced post-operative nausea and vomiting) have led to recommendations for its use. Furthermore, adverse events associated with lidocaine in continuous infusion are minimal.

Based on the early Comfort using Analgesia (eCASH), minimal Sedative and maximal Human care) concepts, the recent PADIS (Pain, Agitation, Delirium, Immobility, Sleep deprivation) recommendations, which determine levels of evidence and research avenues for improving the quality of care, conclude that intravenous lidocaine may be beneficial, but there is a lack of data.

The investigators are therefore proposing a randomised placebo-controlled clinical trial to assess the effectiveness of lidocaine infused continuously for 48 hours on the perceived comfort of post-operative critical care patients, as assessed by the IPREA score.

IPREA, an 18-item score exploring PADIS, is a direct, relevant, objective and reproducible assessment criterion for evaluating algorithms for improving the quality of care. The data on sources of discomfort reveal the importance of pain, dyspnoea, thirst and sleep deprivation, which are all influenced by the analgesia-sedation protocol. Incorporating lidocaine with anti-hyperalgesic properties into the protocol should reduce discomfort in critical care patients.

DETAILED DESCRIPTION:
The choice of analgesia protocol will be left to the discretion of the clinician between MORPHINE CHLORHYDRATE, SUFENTANIL and REMIFENTANIL for objectives of Behavioral Pain Scale (BPS) (3 to 5) or pain visual analogue scale (VAS) < 4.

The use of co-analgesics intraoperatively (Paracetamol, Nefopam, NSAIDs (nonsteroidal anti-inflammatory drugs) such as Ketoprofen or Ibuprofen, Ketamine) is authorised (data not collected).

If a hypnotic is required intraoperatively, the choice of agent is left to the discretion of the clinician.

Once the sedation-analgesia protocol has been discontinued, pain relief is left to the clinician's discretion.

Patients are monitored from randomisation until discharge from the critical care unit or until a maximum of 30 days post-operatively.

In the event of an adverse reaction linked to lidocaine (see list in § 8.2.), the doctor stops administration of the product.

The blind is lifted (see § 9.2 'Insu (or blinding)'). If the patient is in the lidocaine group, the lidocaine plasma concentration is measured to check for a toxic plasma concentration (see § 5.6 'Management of biological samples').

It should be noted that the completion of an assay or discontinuation of treatment does not result in the patient's withdrawal from the clinical trial. Patient follow-up continues until the end of the trial.

If the patient is discharged from critical care before the 30th post-operative day, the patient's vital status on the 30th post-operative day will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18
2. Patient admitted immediately post-operatively in critical care (scheduled or emergency admission, e.g. post-operative exploratory laparotomy, cardiac surgery, major orthopaedic surgery such as polytrauma patients, vascular surgery at risk of complications such as open aortic surgery)
3. Anticipated length of stay in critical care ≥ 48h
4. Membership of a social security scheme
5. Informed consent signed by the patient or by a close relative or legal representative or, failing this, the emergency procedure

Non-inclusion Criteria:

1. Weight over 100 kg
2. Hypersensitivity to one of the active substances used for anaesthesia or to one of the excipients.
3. Known acute porphyria,
4. Pregnant or breast-feeding women
5. Patients who have received or are about to receive peri-medullary analgesia intra-operatively or post-operatively.
6. Patient who has received or will receive loco-regional analgesia intra-operatively or post-operatively.
7. Severe head injury, open cephalic neurosurgery, interventional neuroradiology
8. Recovered cardiorespiratory arrest
9. Noradrenaline doses > 0.5 μg/kg/min
10. Stage IV/V chronic renal failure, not on dialysis
11. Severe hepatocellular insufficiency at inclusion (Child-Pugh C)
12. Bradycardia < 50 bpm on antiarrhythmic drugs
13. Clinical convulsive seizure at inclusion
14. Predictable inability to answer the questionnaire (cognitive impairment, non-Francophone)
15. Known participation in another interventional research study (RIPH1 or RIPH2)
16. Known situation of deprivation of liberty or legal protection (safeguard of justice, guardianship or curatorship)

Exclusion Criteria:

Patients under court protection will be excluded as soon as the investigator is aware of their status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
IPREA | Within 24 hours of discharge from critical care or, failing that, within 24 hours of the 15th day of hospitalisation in critical care.
  Overall score on the Inconforts of Patients in Intensive Care (IPREA) questionnaire.
  Comfort is assessed by the patient him/herself, using a self-assessment scale IPREA, which is explained and conducted with the medical or paramedical staff in the intensive care unit or intensive care unit.
  The IPREA questionnaire was developed specifically for critical incare patients.
  The patient rates his discomfort on a 100 mm graduated visual scale presented horizontally (0: no discomfort, 100: maximum discomfort) for 18 items including (noise, excess light, discomfort of sleeping in intensive care bed, lack of sleep, thirst, hunger, cold, heat, pain, presence of pipes, lack of privacy, anxiety, isolation, limitation of visits, absence of telephone, lack of information, difficulty breathing, depression).
  The overall score is calculated from the average of each item, giving a score from 0 (minimum discomfort) to 100 (maximum discomfort).

SECONDARY OUTCOMES:
IPREA - Sensitivity analysis of the main criterion | Within 24 hours of discharge from critical care or, failing that, within 24 hours of the 15th day of hospitalisation in critical care.
  Sensitivity analysis of the main criterion
  Data from patients who died will be imputed according to the following strategy:
  * the values of patients who died before D7 at the worst value of the IPREA score (100),
  * values for patients who died after D7 by multiple imputation.
  The IPREA questionnaire was developed specifically for critical incare patients. The patient rates his discomfort on a 100 mm graduated visual scale presented horizontally (0: no discomfort, 100: maximum discomfort) for 18 items including (noise, excess light, discomfort of sleeping in intensive care bed, lack of sleep, thirst, hunger, cold, heat, pain, presence of pipes, lack of privacy, anxiety, isolation, limitation of visits, absence of telephone, lack of information, difficulty breathing, depression). The overall score is calculated from the average of each item, giving a score from 0 (minimum discomfort) to 100 (maximum discomfort).
IPREA | Within 24 hours of discharge from critical care or, failing that, within 24 hours of the 7th day of hospitalisation in critical care
  Patients who have died will be considered as not evaluable.
  Overall score on the IPREA questionnaire. Comfort is assessed by the patient him/herself, using a self-assessment scale IPREA, which is explained and conducted with the medical or paramedical staff in the intensive care unit or intensive care unit. The IPREA questionnaire was developed specifically for critical incare patients. The patient rates his discomfort on a 100 mm graduated visual scale presented horizontally (0: no discomfort, 100: maximum discomfort) for 18 items including (noise, excess light, discomfort of sleeping in intensive care bed, lack of sleep, thirst, hunger, cold, heat, pain, presence of pipes, lack of privacy, anxiety, isolation, limitation of visits, absence of telephone, lack of information, difficulty breathing, depression). The overall score is calculated from the average of each item, giving a score from 0 (minimum discomfort) to 100 (maximum discomfort).
IPREA - 8 items | Within 24 hours of discharge from critical care or, failing that, within 24 hours of the 15th day of hospitalisation in critical care.
  Result per item of 8 items of the IPREA score, achieved :
  * Noise
  * Thirst
  * Pain
  * Medical devices (catheters, intubation tubes, etc.)
  * Sleepiness
  * Dyspnoea
  * Anxiety
  * Depression
  Patients who have died will be considered as not evaluable.
  Overall score on the IPREA (Inconforts of Patients in Intensive Care) questionnaire. Comfort is assessed by the patient him/herself, using a self-assessment scale IPREA, which is explained and conducted with the medical or paramedical staff in the intensive care unit or intensive care unit. The IPREA questionnaire was developed specifically for critical incare patients. The patient rates his discomfort on a 100 mm graduated visual scale presented horizontally (0: no discomfort, 100: maximum discomfort) for 18 items. The overall score is calculated from the average of each item, giving a score from 0 (minimum discomfort) to 100 (maximum discomfort).
Cumulative opioid consumption | Over the first 6 post-surgery days
  Cumulative opioid consumption (in mg IV morphine equivalent, or µg Remifentanil or µg Sufentanil)
  In the event of death or premature exit, the criterion will be assessed for the period preceding death or exit.
Duration of invasive mechanical ventilation | Until discharge from critical care, including, in the event of transfer, the stay in critical care in the transfer hospital, or, failing this, until day 30
  Duration of invasive mechanical ventilation in critical care
  In the event of death or premature exit, the criterion will be assessed for the period preceding death or exit.
Occurrence of re-intubation | Within 48 hours of extubation (until discharge from critical care, including, in the event of transfer, the stay in critical care in the transfer hospital, or, failing that, until day 30)
  Occurrence of re-intubation
  In the event of death or premature exit, the criterion will be assessed for the period preceding death or exit.
Duration of sedation | Until discharge from critical care, including, in the event of transfer, the stay in critical care in the transfer hospital, or, failing this, until day 30
  Duration of sedation
  In the event of death or premature exit, the criterion will be assessed for the period preceding death or exit.
Duration of stay in critical care | Until day 30
  Duration of stay in critical care, including, in the event of transfer, the stay in critical care in the transfer hospital
  In the event of death or premature exit, the criterion will be assessed for the period preceding death or exit.
Duration of stay in hospital | Until day 30
  Duration of stay in hospital including, in the event of transfer, the stay in the transfer hospital
  In the event of death or premature exit, the criterion will be assessed for the period preceding death or exit.
Occurrence of pneumonia | During the stay in critical care, including, in the event of transfer, the stay in critical care in the transfer hospital, up to day 30
  Occurrence of pneumonia according to the Recommandations Formalisées d'Experts (RFE) Société française d'anesthésie et de réanimation (SFAR)/Société de Réanimation de Langue Française (SRLF) 2017 'Healthcare-associated pneumonia' criteria in the appendix.
  In the event of death or premature exit, the criterion will be assessed for the period preceding death or exit.
Vital status | Day 30
  Vital status In the event of premature discharge, the vital status will be censored on the date of discharge.
Incidence of serious adverse reactions attributable to lidocaine | For the duration of the treatment and 24 hours after the end of the treatment
  Incidence of serious adverse reactions attributable to lidocaine :
  * Conduction disorders on Electrocardiogram (ECG) not present before treatment,
  * Cardiac arrest
  * Respiratory arrest
  * Anaphylactic shock of any grade
  * Hypotension requiring the introduction of noradrenaline or a significant (>20%) increase in the dose of noradrenaline (if treatment with noradrenaline was already underway when the experimental treatment was initiated).
  * Bradycardia requiring the introduction of atropine
  * Bradycardia requiring the introduction of dobutamine
  * Bradycardia requiring the introduction of isoprenaline
  * Convulsive seizures
  * Presumed lidocaine intoxication defined by the presence of two of the following:
  * Vertigo
  * Dysgeusia
  * Perioral and lingual paresthesias, dysarthria
  * Blurred vision
  * Tinnitus, hearing dysfunction
  * Tremor
  In the event of death or premature exit, the criterion will be assessed for the period preceding death or exit.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie MASSERET, MD, Principal Investigator — Rennes University Hospital
Locations (15):
- France (15):
  - CHU d'Angers - RCA (Réanimation Chirurgicale A), Angers
  - CHU d'Angers - RCB (Réanimation Chirurgicale B), Angers
  - CHU de Brest - Réanimation Cardiaque, Brest
  - CH Louis Pasteur (Chartres) - Réanimation, Chartres
  - CHU de Nantes - Hôpital Guillaume et René Laennec - Réanimation Chirurgicale Polyvalente, Nantes
  - CHU de Nantes - Hôpital Guillaume et René Laennec - Réanimation CTCV, Nantes
  - CHU de Nantes - Hôtel-Dieu - Réanimation chirurgicale, Nantes
  - CHU de Poitiers - Réanimation Chirurgicale, Poitiers
  - CHU de Rennes - Réanimation chirurgicale, Rennes
  - CHU de Rennes - Réanimation CTCV, Rennes
  - CH de Saint-Nazaire - Réanimation médico-chirurgicale - Unité de Surveillance Continue (USC), Saint-Nazaire
  - CHRU de Tours - Hôpital Trousseau - Réanimation Chirurgicale, Tours
  - CHRU de Tours - Hôpital Trousseau - Réanimation URTC, Tours
  - CHRU de Tours - Hôpital Trousseau - Unité de Soins Continus, Tours
  - CH Bretagne Atlantique (Vannes) - Réanimation - Unité de Surveillance Continue, Vannes

IPD SHARING:
Plan to Share IPD: No